CLINICAL TRIAL: NCT01376830
Title: Biomarkers and Clinical Characteristics That Identify the Risk of an Exacerbation Following Viral Upper Respiratory Tract Infections in COPD Patients
Brief Title: Characteristics That Identify Exacerbation Risk Following Colds in COPD Patients
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: CRO1697
Record Dates: First submitted 2011-06-17; First posted 2011-06-20 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Exacerbations; Viruses
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum,nasal lavage, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients

SUMMARY:
Respiratory virus infections are a common cause of COPD exacerbations and antiviral therapies have potential as treatments for exacerbations. However it is likely that treating patients when they present with an exacerbation with antiviral drugs will be too late to be effective and earlier treatment at the time of the initial upper respiratory tract infection (URTI) will be required. The incidence of exacerbations following URTIs in COPD patients, and whether there are host factors and biomarkers that can identify the risk of this, is unknown. The aims of this study are to establish the proportion of viral URTIs that progress to an acute exacerbation in COPD patients and identify clinical, viral and biological markers that predict risk of an exacerbation following an URTI. In addition we will determine the frequency of, and risk factors for, bacterial infection following viral URTIs in COPD patients. This data will permit development of a model combining baseline patient characteristics, clinical measurements and biomarkers to predict exacerbation risk following viral URTI in COPD patients. The results will open the way for trials of antiviral therapy in COPD exacerbations and targeting of treatment to high risk patients.

DETAILED DESCRIPTION:
Research Protocol

Biomarkers and clinical characteristics that identify the risk of an exacerbation following viral upper respiratory tract infections in COPD patients

Chief Investigator: Dr Patrick Mallia Co-investigators: Professor Sebastian Johnston Dr Sarah Elkin

Study Site The study will take place at St Mary's Hospital, London - part of the Imperial College Healthcare NHS Trust.

1. Background COPD exacerbations are a major cause of health care costs, morbidity and mortality. Current therapies are only partially effective and have considerable side effects so new treatments are urgently needed. 40 - 50% of COPD exacerbations are associated with virus infections and the commonest viruses detected are rhinoviruses and influenza1,2. Sensitive and rapid diagnostic techniques for viral infections have recently become available3 and drugs effective against rhinovirus and influenza have been developed4, making antiviral therapy a realistic potential treatment option for COPD exacerbations. However our understanding of the relationship between viral infections and COPD exacerbations remains limited and a more information is required before trials of antiviral therapies are carried out.

An experimental model of COPD exacerbation We have developed a model of COPD exacerbation using experimental rhinovirus infection in COPD patients that allows us to study a number of outcomes in a carefully controlled manner not possible with naturally occurring infections5,6. This model has provided novel data regarding the relationships between virus infection and exacerbations. Following rhinovirus infection subjects developed symptoms of upper respiratory tract infection (URTI) that commenced on day 2 post-inoculation and peaked on day 4, followed by the typical lower respiratory tract symptoms of an acute exacerbation that commenced on day 5 and peaked on day 9. Airflow obstruction and lower airways inflammation also peaked on day 9. Maximum virus load occurred on day 4 in nasal lavage and day 5 in sputum. In naturally occurring exacerbations patients present 3-4 days after the onset of exacerbation symptoms7 and our data shows that the peak of virus replication is likely to have already occurred by this time. Therefore intervention with antiviral drugs at the time of exacerbation may be too late. 63% of COPD subjects in our study developed bacterial infections following experimental rhinovirus infection. While virus load peaked on day 5 most bacterial infections occurred later on days 12 and 15 post-inoculation, suggesting that rhinovirus infection increases susceptibility to bacterial infection. Therefore treatment of viral infections may have the additional benefit of reducing secondary bacterial infections.

Predicting risk of exacerbation: preliminary data from the experimental model Data obtained from our experimental model allowed us to evaluate relationships between markers at the time of initial URTI and measures of subsequent exacerbation severity. Peak upper respiratory symptoms correlated with peak lower respiratory scores (p=0.0037, r=0.58), sputum inflammatory cells counts (p=0.018, r=0.5) and sputum virus load (p=0.014, r=0.51). The fall in peak expiratory flow on day 5 correlated with peak lower respiratory scores (p=0.023, r=-0.47), breathlessness scores (p=0.0079, r=-0.54) and sputum virus load (p=0.03, r=-0.45). Blood neutrophils on day 5 correlated with peak fall in FEV1 (p=0.0072, r=-0.55), total leukocyte count on day 5 with peak fall in FEV1/FVC (p=0.04, r=-0.43) and nasal lavage virus load on day 5 correlated with peak fall in FEV1 (p=0.0186, r=-0.49). These data suggest that parameters such as symptoms, airflow obstruction, peripheral leukocyte counts and virus load measured during an URTI in COPD patients correlate with subsequent lower respiratory symptoms, airflow obstruction and airways inflammation and could predict the risk of exacerbation. However this study was in a small number of patients with mild-moderate COPD and these findings need to be explored in a larger cohort of patients with a wider range of COPD severity with naturally-occurring infections.

Biomarkers Exacerbations are defined by increases in symptoms and the diagnosis depends on a subjective assessment of symptoms by patients and health care providers. No markers - either biological or physiological - exist that can be used to define an exacerbation. Exacerbations are associated with airways inflammation but direct measurement of inflammatory markers is difficult as bronchoalveolar lavage and endobronchial biopsy are too invasive, and sputum and exhaled breath condensate too complex and time-consuming to be practical in routine clinical practice. Blood is easily obtainable for measurement of biomarkers but it is not established that systemic markers reflect airways inflammation or correlate with clinical outcomes in COPD exacerbations. Nasal samples are also easy to obtain and there is data showing nasal inflammatory markers correlate with lower airway inflammation8 and we have reported that IL-8 and IL-6 are elevated in nasal lavage following experimental rhinovirus infection5. A number of biomarkers have been investigated both as markers of COPD exacerbations and indicators of specific aetiologies. Copeptin9 and serum amyloid A (SAA)10 correlate with clinical outcomes in COPD exacerbations, interferon-induced protein-10 (IP-10)11 and neopterin have been identified as potential markers of viral respiratory infections12,13 and procalcitonin as a marker of bacterial infection14. However none of these markers have been investigated specifically as predictors of outcomes following URTI in COPD.

Relationship between viral URTI and COPD exacerbations Data from our study suggests that treatment at the time of the initial URTI may be required to prevent virus-induced exacerbations. However this strategy risks treating URTIs that do not progress to an exacerbation resulting in over-treatment. Only one study has examined exacerbations following URTIs in COPD patients and found 43% of URTIs were followed by exacerbations15. However in this study URTIs were identified retrospectively from symptom diary cards and therefore it was not proven that the symptoms were caused by viral infection. Up to 75% of COPD patients complain of upper respiratory symptoms when clinically stable16 so upper respiratory symptoms caused by factors other than viral infections would have weakened the association between URTI and COPD exacerbations in this study. The true association is likely to be higher and can only be determined by virological confirmation of infection. Also the risk of exacerbation following a viral URTI may not be the same for all COPD patients but may be influenced by host factors such as FEV1, previous exacerbation history and smoking status. Currently no data is available regarding how these factors may influence risk of exacerbation following a viral URTI. All studies to date of COPD exacerbations have recruited patients when they present with symptoms of an exacerbation. Therefore the opportunity to investigate the relationship between a preceding URTI and the exacerbation has been missed. The aim of this study is to recruit a cohort of COPD patients and investigate them when they develop an URTI so that the relationship with a subsequent exacerbation can be examined in a prospective manner.

2) Study Aims

1. To establish the proportion of URTIs with a confirmed viral aetiology in COPD patients that progress to an acute exacerbation and determine the specific viral aetiologies.
2. To identify clinical, viral and biological markers that predict progression of an URTI to an exacerbation and correlate with exacerbation severity.
3. To determine baseline clinical characteristics that identify patients at high risk of developing exacerbations following a viral URTI.
4. To determine the frequency of, and risk factors for, bacterial infection following viral URTI in COPD patients.
5. To develop a model combining baseline patient characteristics, clinical measurements and biomarkers that will predict exacerbation risk following viral URTI in COPD patients.

3) Methods Study subjects A cohort of 100 COPD subjects will be recruited from the Chest and Allergy clinic at St Mary's Hospital, Paddington part of Imperial College Healthcare NHS Trust and community clinics within the local areas of Westminster and Kensington and Chelsea.

Inclusion Criteria The principal inclusion criterion is patients who are 40-85 years old with a diagnosis of COPD confirmed with spirometry.

Exclusion Criteria

* Participants who have difficulty understanding English so would not be able to answer symptom questionnaires.
* Participants who have another medical condition such as advanced cancer that means they have a life expectancy less than 2 years and so would not be able to complete follow-up.
* Participants who would find it difficult to attend for frequent visits to hospital will also be excluded.

Baseline visit Following informed consent participants will have a baseline visit at which they will have detailed clinical characterisation including documentation of smoking status, co-morbidities, exacerbation frequency and medications and measurement of lung function (FEV1, FVC, FEV1,/FVC, PEF, transfer coefficient). Sputum, nasal fluid and blood will be collected for baseline assessment of bacterial and viral colonisation and measurement of airways inflammation and biomarkers. During the course of the study the participants will have repeat visits with the same assessment and sampling carried out every 3 months. The purpose of this is to document any changes in clinical status (e.g. change in smoking status) and to ensure that if a cold/exacerbation occurs there will be a stable visit with which to compare parameters within the last 3 months.

Following the baseline visit the participants will commence a record of lower respiratory symptoms using the Exacerbations of Chronic Pulmonary Disease Tool (EXACT), a new patient-reported outcome diary that has been validated in COPD cohort studies17. They will continue their usual medications and medical care but will be advised to contact the investigators if they develop symptoms of a cold or an exacerbation. They will be contacted by telephone weekly in an attempt to identify all episodes of increased respiratory symptoms.

Cold visit Subjects will be advised to report to the investigators if they develop symptoms of an URTI. When this occurs they will be seen within 24 hours for a 'cold visit' - the details of this visit are shown below.

URTI symptoms will be quantified using the Wisconsin Upper Respiratory Symptom Survey (WURSS-21)18 questionnaire. The WURSS-21 is a quality of life assessment that measures the health-related effects of the common cold and has been used to predict exacerbations following URTI in asthmatics19. To obtain WURSS-21 scores in COPD subjects without a cold a subgroup of stable subjects will be administered the WURSS-21 for 14 consecutive days. FEV1, FVC, FEV1,/FVC and PEF will be measured and samples of nasal fluid, induced sputum and blood collected.

All subjects will be seen 7 days after the cold visit with repeat sampling unless they develop an exacerbation prior to this. As exacerbations are defined by symptoms and symptom perception is subjective the purpose of this visit will be to measure objective markers such as lung function and inflammatory markers in the clinical samples collected. Comparing these between participants who do and do not report exacerbations will provide more objective evidence that an exacerbation has occurred in addition to symptoms.

Exacerbation visit When subjects develop an URTI they will monitored for symptoms of a subsequent exacerbation and if this occurs they will have a further visit termed the 'exacerbation visit'. If participants develop an exacerbation without a preceding URTI they will also be seen. Clinical assessment including physical examination, symptom scores and spirometry will be carried out to evaluate exacerbation severity and the same clinical samples as the cold visit collected. Subjects will have further visits 2 and 6 weeks after exacerbation onset with repeat assessment and clinical sampling.

Milestones COPD patients have an average of 1-2 colds per year so recruiting a cohort of 100 subjects and following them for 24 months to include 4 seasons of peak rhinovirus activity should provide at least 200 episodes of URTI to evaluate. We will then require 6 months to complete the laboratory analyses and analyse the data.

4) Study Procedures Throat swab A sterile dry cotton-headed swab is used to obtain samples from the pharynx for virus detection. This is performed with the subject sitting. Ensure adequate lighting and use a tongue depressor if required. Remove the swab from the container carefully to ensure the tip is not contaminated, and swab the dorsal aspect of the pharynx and soft palate, avoiding the tongue. Place swab into a dry container and freeze at -80°C prior to analysis and another into bacteriology culture medium.

Nasosorption

Nasal lining fluid will be collected using the Synthetic Absorptive Matrix (SAM) method. Fluid volumes of 50-100μL are obtained and 50μL is enough to measure up to 20 analytes using the MSD platform (http://www.meso-scale.com), which we have already used to assay soluble mediators in human studies and custom made plates to measure selected mediators can be obtained. Strips of SAM will be used for 2 minutes in the nostril to obtain repeated samples of neat nasal ELF. This is a painless minimally invasive procedure that will not require any local anaesthetic. Following sampling, SAM will be placed in a 1mL microfuge spin filter tube containing 100μL of elution buffer (PBS/1% bovine serum albumin/1% Triton®). In order to determine the volume of fluid obtained by nasosorption and hence the final concentration of soluble mediators in ELF, the weight of the SAM before and after sampling must be known. The following procedure must be followed:

* Record the dry weight of the SAM (DS)
* Record the dry empty weight of the microfuge tube (DT)
* Record the combined weight of the microfuge tube containing SAM in elution buffer (CW)
* Calculate and record weight of ELF (mg):

Weight of ELF = CW - (DT + DS + 100) (100mg is the weight of 100μL of elution buffer) The SAM will be transported on dry ice to the laboratory.

Nasal Lavage

Nasal lavage is performed using the following technique:

* Procedure to occur in negative-pressure room on ICRRU
* 5mL of 0.9% saline is introduced into one nostril using a syringe with the subject sitting with the head tilted back.
* The saline is held in the nose for 5 seconds then blown into a sterile pot. The procedure is then repeated for the other nostril.
* The fluid is then aliquotted into sterile microfuge tubes and centrifuged for analysis of cells and supernatants are frozen at -80°C.

Nasal lavage fluid will be analysed with PCR for respiratory viruses. Any samples that are positive for rhinovirus will be further analysed with a quantitative PCR to determine the virus load.

Blood sampling Blood will be taken at the baseline visit for separation of serum for measurement of inflammatory markers and measurement of C-reactive protein and a full blood count. These will be processed in the Respiratory Medicine laboratories in the Medical School Building, St Mary's Campus.

The total amount of blood taken at each visit would amount to 20mL.

Induced Sputum Sputum will be induced and processed using standard protocols20. Briefly participants will be pre-medicated with 200mg salbutamol via metered dose inhaler and large volume spacer and baseline FEV1 measured. 3% saline will be administered with a DeVilbiss UltraNeb99 ultrasonic nebuliser in 2 minute periods and FEV1 measured again. If FEV1 falls by 20% the procedure will be discontinued and further salbutamol administered. Otherwise the procedure will be continued and FEV1 measured every 2 minutes until an adequate sputum sample is obtained. Sputum will be processed within 2 hours of induction. Sputum plugs will be selected from saliva by macroscopic inspection of the sample and an aliquot selected and stored unprocessed at -80oC for qRT-PCR for virus detection. An aliquot of sputum will also be kept for bacterial detection. The remaining sample will be weighed, 0.1% Dithiothreitol (DTT) added in the ratio 4ml DTT to 1g sputum and the mixture agitated and filtered. The same volume PBS added, the filtrate centrifuged and the supernatant aliquotted and stored at -80°C. The cell pellet will be washed and resuspended and the cells counted to obtain total cell counts. Cytospins will be prepared and stained using Shandon Diffquick kit (Thermo Shandon Ltd, Cheshire, UK), coded and counted blind to study status to obtain differential cell counts. Cell counts will be expressed as a percentage of at least 400 inflammatory cells.

5) Regulatory issues Ethics approval Approval has been obtained from the East London Research Ethics Committee for this study. The study will be submitted for Site Specific Assessment (SSA) at Imperial College Healthcare NHS Trust. The Chief Investigator will require a copy of the R&D approval letter before accepting participants into the study. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Declaration of Helsinki 1964 and later revisions.

Consent Consent to enter the study will be sought from each participant only after a full explanation has been given, an information leaflet offered, time allowed for consideration, and any questions participants may have answered. Signed participant consent will be obtained. The right of the participant to refuse to participate without giving reasons must be respected. After the participant has entered the study the clinician remains free to give alternative treatment to that specified in the protocol at any stage if he/she feels it is in the participant's best interest, but the reasons for doing so should be recorded. In these cases the participants remain within the study for the purposes of follow-up and data analysis. All participants are free to withdraw at any time from the protocol treatment without giving reasons and without prejudicing further treatment.

Confidentiality The Chief Investigator and all of the research team will preserve the confidentiality of participants taking part in the study and abide by the Data Protection Act.

Indemnity Imperial College, London as sponsor of this study holds negligent and non-negligent harm insurance policies which apply to this study. These have been arranged through the Joint Research Office.

Sponsor Imperial College London will act as the main sponsor for this study. Delegated responsibilities will be assigned to the NHS trust taking part in this study.

Funding Following a successful application to the Biomedical Research Centre (BRC) of the Imperial Healthcare NHS Trust and Imperial College the BRC is funding this study. The investigators will not receive any additional payment above their normal salaries. Participants in the study will have their travel costs refunded.

Audits and inspections The study may be subject to inspection and audit by Imperial College London under their remit as sponsor and other regulatory bodies to ensure adherence to GCP and the NHS Research Governance Framework for Health and Social Care (2nd edition).

Study Management The day-to-day management of the study will be co-ordinated by Dr Patrick Mallia, Chief Investigator for the project.

Publication Policy Our expectation is that after analysis the data from this study will be widely distributed in the medical and scientific community. Facilitated with presentations at local, national and international meetings, we hope to publish widely in the medical literature. In addition we have an excellent media department at Imperial College and publicise research that has public interest when it is published. No identifying participant information will be published.

6) Adverse Events Definitions Adverse Event (AE): any untoward medical occurrence in a patient or clinical study subject.

Serious Adverse Event (SAE): any untoward and unexpected medical occurrence or effect that:

* Results in death
* Is life-threatening - refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe
* Requires hospitalisation
* Results in persistent or significant disability or incapacity
* Is a congenital anomaly or birth defect

Reporting procedures All adverse events should be reported. Depending on the nature of the event the reporting procedures below should be followed. Any questions concerning adverse event reporting should be directed to the Chief Investigator in the first instance.

Non serious AEs All such events, whether expected or not, should be recorded.

Serious AEs An SAE form should be completed and faxed to the Chief Investigator and the Sponsor within 24 hours.

All SAEs should be reported to the East London Research Ethics Committee where in the opinion of the Chief Investigator, the event was:

* 'related', i.e. resulted from the administration of any of the research procedures; and
* 'unexpected', i.e. an event that is not listed in the protocol as an expected occurrence

Reports of related and unexpected SAEs should be submitted to ethics, the sponsor and the R&D office within 15 days of the Chief Investigator becoming aware of the event, using the NRES SAE form for non-IMP studies.

Contact details for reporting SAEs Fax: 020 7262 8913 for the attention of Dr Patrick Mallia Tel: 020 7594 3751 (Mon to Fri 09.00 - 17.00)

7) Track Records Our group has an established record of high quality research in the field of viral infections in asthma and COPD. We have established protocols for PCR detection of respiratory viruses, quantitative PCR for rhinovirus and have collaborated with Imperial College Healthcare NHS Trust Microbiology Laboratory for semi-quantitative bacterial cultures. We have established protocols and experience in measuring inflammatory mediators in nasal fluid and sputum supernatants and are developing expertise in use of the MSD platform. Dr Elkin has experience in recruiting cohorts of COPD patients for longitudinal clinical trials.

8) Expected impact This study will be the first to determine the relationship between viral URTI and exacerbations in COPD patients. It will establish clinical factors and biomarkers that predict the risk of an exacerbation following an URTI. The data obtained will be of enormous interest to the pharmaceutical industry and clinical researchers as it will open the way for trials of antiviral therapies for virus-induced COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Age 40-85

Exclusion Criteria:

* Unable to understand English
* Expected life expectancy < 2 years
* Unable to attend hospital

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of colds followed by exacerbations in COPD patients | 2 years

SECONDARY OUTCOMES:
Clinical characteristics that identify high risk of exacerbation following a cold in COPD patients | 2 years
Biomarkers that identify the risk of exacerbation following colds in COPD patients | 2 years
Changes in bacterial flora following colds in COPD patients | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mallia, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

REFERENCES:
- [Background] Seemungal T, Harper-Owen R, Bhowmik A, Moric I, Sanderson G, Message S, Maccallum P, Meade TW, Jeffries DJ, Johnston SL, Wedzicha JA. Respiratory viruses, symptoms, and inflammatory markers in acute exacerbations and stable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1618-23. doi: 10.1164/ajrccm.164.9.2105011. PMID 11719299
- [Background] Papi A, Bellettato CM, Braccioni F, Romagnoli M, Casolari P, Caramori G, Fabbri LM, Johnston SL. Infections and airway inflammation in chronic obstructive pulmonary disease severe exacerbations. Am J Respir Crit Care Med. 2006 May 15;173(10):1114-21. doi: 10.1164/rccm.200506-859OC. Epub 2006 Feb 16. PMID 16484677
- [Background] Do DH, Laus S, Leber A, Marcon MJ, Jordan JA, Martin JM, Wadowsky RM. A one-step, real-time PCR assay for rapid detection of rhinovirus. J Mol Diagn. 2010 Jan;12(1):102-8. doi: 10.2353/jmoldx.2010.090071. Epub 2009 Nov 30. PMID 19948820
- [Background] Hayden FG, Herrington DT, Coats TL, Kim K, Cooper EC, Villano SA, Liu S, Hudson S, Pevear DC, Collett M, McKinlay M; Pleconaril Respiratory Infection Study Group. Efficacy and safety of oral pleconaril for treatment of colds due to picornaviruses in adults: results of 2 double-blind, randomized, placebo-controlled trials. Clin Infect Dis. 2003 Jun 15;36(12):1523-32. doi: 10.1086/375069. Epub 2003 Jun 6. PMID 12802751
- [Background] Mallia P, Message SD, Kebadze T, Parker HL, Kon OM, Johnston SL. An experimental model of rhinovirus induced chronic obstructive pulmonary disease exacerbations: a pilot study. Respir Res. 2006 Sep 6;7(1):116. doi: 10.1186/1465-9921-7-116. PMID 16956406
- [Background] Mallia P, Message SD, Gielen V, Contoli M, Gray K, Kebadze T, Aniscenko J, Laza-Stanca V, Edwards MR, Slater L, Papi A, Stanciu LA, Kon OM, Johnson M, Johnston SL. Experimental rhinovirus infection as a human model of chronic obstructive pulmonary disease exacerbation. Am J Respir Crit Care Med. 2011 Mar 15;183(6):734-42. doi: 10.1164/rccm.201006-0833OC. Epub 2010 Oct 1. PMID 20889904
- [Background] Wilkinson TM, Donaldson GC, Hurst JR, Seemungal TA, Wedzicha JA. Early therapy improves outcomes of exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1298-303. doi: 10.1164/rccm.200310-1443OC. Epub 2004 Feb 27. PMID 14990395
- [Background] Hurst JR, Donaldson GC, Perera WR, Wilkinson TM, Bilello JA, Hagan GW, Vessey RS, Wedzicha JA. Use of plasma biomarkers at exacerbation of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Oct 15;174(8):867-74. doi: 10.1164/rccm.200604-506OC. Epub 2006 Jun 23. PMID 16799074
- [Background] Stolz D, Christ-Crain M, Morgenthaler NG, Leuppi J, Miedinger D, Bingisser R, Muller C, Struck J, Muller B, Tamm M. Copeptin, C-reactive protein, and procalcitonin as prognostic biomarkers in acute exacerbation of COPD. Chest. 2007 Apr;131(4):1058-67. doi: 10.1378/chest.06-2336. PMID 17426210
- [Background] Bozinovski S, Hutchinson A, Thompson M, Macgregor L, Black J, Giannakis E, Karlsson AS, Silvestrini R, Smallwood D, Vlahos R, Irving LB, Anderson GP. Serum amyloid a is a biomarker of acute exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Feb 1;177(3):269-78. doi: 10.1164/rccm.200705-678OC. Epub 2007 Nov 15. PMID 18006888
- [Background] Quint JK, Donaldson GC, Goldring JJ, Baghai-Ravary R, Hurst JR, Wedzicha JA. Serum IP-10 as a biomarker of human rhinovirus infection at exacerbation of COPD. Chest. 2010 Apr;137(4):812-22. doi: 10.1378/chest.09-1541. Epub 2009 Oct 16. PMID 19837822
- [Background] Ip M, Rainer TH, Lee N, Chan C, Chau SS, Leung W, Leung MF, Tam TK, Antonio GE, Lui G, Lau TK, Hui DS, Fuchs D, Renneberg R, Chan PK. Value of serum procalcitonin, neopterin, and C-reactive protein in differentiating bacterial from viral etiologies in patients presenting with lower respiratory tract infections. Diagn Microbiol Infect Dis. 2007 Oct;59(2):131-6. doi: 10.1016/j.diagmicrobio.2007.04.019. Epub 2007 Jul 26. PMID 17662560
- [Background] Rainer TH, Chan CP, Leung MF, Leung W, Ip M, Lee N, Cautherley GW, Graham CA, Fuchs D, Renneberg R. Diagnostic utility of CRP to neopterin ratio in patients with acute respiratory tract infections. J Infect. 2009 Feb;58(2):123-30. doi: 10.1016/j.jinf.2008.11.007. Epub 2008 Dec 13. PMID 19073345
- [Background] Stolz D, Christ-Crain M, Bingisser R, Leuppi J, Miedinger D, Muller C, Huber P, Muller B, Tamm M. Antibiotic treatment of exacerbations of COPD: a randomized, controlled trial comparing procalcitonin-guidance with standard therapy. Chest. 2007 Jan;131(1):9-19. doi: 10.1378/chest.06-1500. PMID 17218551
- [Background] Hurst JR, Donaldson GC, Wilkinson TM, Perera WR, Wedzicha JA. Epidemiological relationships between the common cold and exacerbation frequency in COPD. Eur Respir J. 2005 Nov;26(5):846-52. doi: 10.1183/09031936.05.00043405. PMID 16264045
- [Background] Roberts NJ, Lloyd-Owen SJ, Rapado F, Patel IS, Wilkinson TM, Donaldson GC, Wedzicha JA. Relationship between chronic nasal and respiratory symptoms in patients with COPD. Respir Med. 2003 Aug;97(8):909-14. doi: 10.1016/s0954-6111(03)00114-8. PMID 12924517
- [Background] Leidy NK, Wilcox TK, Jones PW, Roberts L, Powers JH, Sethi S; EXACT-PRO Study Group. Standardizing measurement of chronic obstructive pulmonary disease exacerbations. Reliability and validity of a patient-reported diary. Am J Respir Crit Care Med. 2011 Feb 1;183(3):323-9. doi: 10.1164/rccm.201005-0762OC. Epub 2010 Sep 2. PMID 20813886
- [Background] Barrett B, Brown R, Voland R, Maberry R, Turner R. Relations among questionnaire and laboratory measures of rhinovirus infection. Eur Respir J. 2006 Aug;28(2):358-63. doi: 10.1183/09031936.06.00002606. Epub 2006 Apr 26. PMID 16641127
- [Background] Walter MJ, Castro M, Kunselman SJ, Chinchilli VM, Reno M, Ramkumar TP, Avila PC, Boushey HA, Ameredes BT, Bleecker ER, Calhoun WJ, Cherniack RM, Craig TJ, Denlinger LC, Israel E, Fahy JV, Jarjour NN, Kraft M, Lazarus SC, Lemanske RF Jr, Martin RJ, Peters SP, Ramsdell JW, Sorkness CA, Sutherland ER, Szefler SJ, Wasserman SI, Wechsler ME; National Heart, Lung and Blood Institute's Asthma Clinical Research Network. Predicting worsening asthma control following the common cold. Eur Respir J. 2008 Dec;32(6):1548-54. doi: 10.1183/09031936.00026808. Epub 2008 Sep 3. PMID 18768579
- [Background] Efthimiadis A, Spanevello A, Hamid Q, Kelly MM, Linden M, Louis R, Pizzichini MM, Pizzichini E, Ronchi C, Van Overvel F, Djukanovic R. Methods of sputum processing for cell counts, immunocytochemistry and in situ hybridisation. Eur Respir J Suppl. 2002 Sep;37:19s-23s. doi: 10.1183/09031936.02.00001902. No abstract available. PMID 12361358
- [Derived] Calderazzo MA, Trujillo-Torralbo MB, Finney LJ, Singanayagam A, Bakhsoliani E, Padmanaban V, Kebadze T, Aniscenko J, Elkin SL, Johnston SL, Mallia P. Inflammation and infections in unreported chronic obstructive pulmonary disease exacerbations. Int J Chron Obstruct Pulmon Dis. 2019 Apr 10;14:823-832. doi: 10.2147/COPD.S191946. eCollection 2019. PMID 31114182